CLINICAL TRIAL: NCT00340106
Title: Prevention of Environmental Tobacco Smoke (ETS) Exposure to Children, Ages 0-12 Months
Brief Title: Prevention of Environmental Tobacco Smoke Exposure in Children 0-12 Months Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905211; 05-CH-N211
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-18

CONDITIONS: Environmental Tobacco Smoke (ETS)
Keywords: Infant Health Study; Environmental Tobacco Smoke; Infant Health
MeSH Terms: interventions — Counseling

INTERVENTIONS:
Behavioral: Counseling

SUMMARY:
This study will: 1) test the effectiveness of a program to prevent the exposure of infants to environmental tobacco smoke; and 2) evaluate the health effects associated with prenatal and postpartum exposure to tobacco smoke products and environmental tobacco smoke among infants.

African-American and Hispanic women who are 18 years of age or older, and who are between 28 and 35 weeks pregnant may be eligible for this study. Participants complete an interview and home visit assessment and are then randomly assigned to participate in Program A or Program B of the study, as follows:

Program A: Involves discussions with an Infant Health Advisor about parenting skills to promote child safety and infant growth and development, such as ways to prevent childhood injuries caused by falls, poisons, and other hazards.

Program B: Involves discussions with an Infant Health Advisor about ways to prevent infant tobacco smoke exposure, such as how to adopt smoke-free household rules in the home and how to work with friends and family members to prevent the baby from being exposed to tobacco smoke. In addition, participants who smoked cigarettes before becoming pregnant or while pregnant are given advice on how to quit smoking and how to remain a non-smoker once the baby is born.

Participants come to the clinic four times- once during a regularly scheduled prenatal visit and again when the baby is 6 weeks, 4 months, and 6 months old - to see the Infant Health Advisor for the activities described above in Program A or Program B. Between visits, the Advisor calls the participant to check on her progress regarding the program objectives. In addition, the study involves the following for all participants:

* Telephone interview during the week after joining the study to obtain information on participant's background, pregnancy and family history, tobacco use and exposure to other people's cigarette smoke during pregnancy, strategies to reduce tobacco use and exposure, stressful life events, drug and alcohol use during pregnancy, and sources of social support. Similar interviews are repeated when the baby is 6 weeks old, and again when the baby is 4 months, 6 months, and 12 months old.
* Home visit about 1 week after entering the study to check the home for possible safety hazards to the baby and to place one or more nicotine air monitors (small plastic objects that measure the amount of tobacco smoke in the air of each room). The home visitor returns a week late...

DETAILED DESCRIPTION:
ETS exposure is a major public health concern, and tobacco use is one of the 10 Healthy People 2010 leading health indicators. Despite the body of evidence showing the adverse effects of in-utero and postnatal exposure to tobacco smoke products (TSP) and environmental tobacco smoke (ETS) to the respiratory health in children, studies continue to be needed to elucidate when TSP exposure causes the greatest damage, possible mechanisms that underlie the damage, and how harm to the respiratory system of infants and vulnerable children can be prevented. and, while some efforts to reduce prenatal and childhood ETS exposure over the past decade have been successful, there is a paucity of randomized, controlled, intervention studies in the literature targeting ETS exposure reduction among infants age 0-12 months. Moreover, the effectiveness of ETS exposure prevention interventions in reducing the occurrence or severity of health symptoms and outcomes has rarely been systematically evaluated.

ELIGIBILITY:
* INCLUSION CRITERIA:

English-speaking women over age 18, who self-identify as African American, Black or Hispanic, live in the DC metropolitan area, and who have a singleton pregnancy will be enrolled in this study.

EXCLUSION CRITERIA:

Exclusionary criteria include women reporting diagnosis of major psychiatric illnesses, current incarceration, or suicidal ideation, or who initiate prenatal care after 28 weeks. At postpartum, women who have lost custody of the child, are in withdrawal from addictive substances requiring hospitalization or methadone treatment will be deemed ineligible to remain in the study. Further, all women who report delivery complications requiring a hospital stay of 7 days or longer or the infants' admissions to the NICU (or NICU step down unit) for more than 12 hours, including infant prematurity less than 34 weeks, or infant birth weight less than 1800gm (i.e. 4.9 pounds) will be considered ineligible to continue in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2005-07-25; Primary Completion 2010-03-05 (Actual); Study Completion 2010-05-18 (Actual)

PRIMARY OUTCOMES:
Infant ETS exposure 1)Maternal reports of infant ETS exposure at home and 2) Infant urinary cotinine levels.

SECONDARY OUTCOMES:
Household ETS exposure levels, and maternal salivary cotinine levels.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GW University Medical Center, Washington D.C., District of Columbia
  - Providence Hospital, Washington D.C., District of Columbia

REFERENCES:
- [Background] Lodrup Carlsen KC, Carlsen KH. Effects of maternal and early tobacco exposure on the development of asthma and airway hyperreactivity. Curr Opin Allergy Clin Immunol. 2001 Apr;1(2):139-43. doi: 10.1097/01.all.0000010998.15560.b6. PMID 11964681
- [Background] Chan-Yeung M, Manfreda J, Dimich-Ward H, Ferguson A, Watson W, Becker A. A randomized controlled study on the effectiveness of a multifaceted intervention program in the primary prevention of asthma in high-risk infants. Arch Pediatr Adolesc Med. 2000 Jul;154(7):657-63. doi: 10.1001/archpedi.154.7.657. PMID 10891016
- [Background] Chilmonczyk BA, Palomaki GE, Knight GJ, Williams J, Haddow JE. An unsuccessful cotinine-assisted intervention strategy to reduce environmental tobacco smoke exposure during infancy. Am J Dis Child. 1992 Mar;146(3):357-60. doi: 10.1001/archpedi.1992.02160150097031. PMID 1543187